CLINICAL TRIAL: NCT06322498
Title: Inflammation Markers in Fluid Aspirate From a Scarred Uterine vs. a Normal Uterine Cavity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Chana Adler, Principal Investigator, IVF clinic physician, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INFLAM.UTERUS-HMO-CTIL
Record Dates: First submitted 2022-07-10; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Infertility Due to Nonimplantation; Infertility Secondary; Cesarean Section Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intact uterus (Experimental): Patients with intact uterus
  Interventions: Diagnostic Test: Uterine lavage
- Scarred uterus (Experimental): Patients with scarred uterus
  Interventions: Diagnostic Test: Uterine lavage

INTERVENTIONS:
Diagnostic Test: Uterine lavage — Infusion of 2ml 0.9%NACL into the uterine cavity and aspiration of the fluid

SUMMARY:
A prospective study that will take place in the hydrosonography clinic, comparing patients with an intact uterus to those who had a caesarean section. Eligible patients will preform a transvaginal ultrasound for evaluation of presence of a niche. After fixation of the transcervical catheter, we will flush 2 ml sterile NaCl 0.9% into the uterine cavity and aspirate the fluid. After collecting all samples, the samples will be snap frozen and stored at -80o C, until they undergo an immunological analysis.

ELIGIBILITY:
Inclusion Criteria:

- Patients suffering from infertility and assigned for a hydrosonography exam for assessment of the integrity of the uterus and fallopian tubes.

Exclusion Criteria:

1. Patients with hydrosalpinx/pyosalpinx/sactosalpinx
2. Patients who went through surgical correction of a niche
3. Hormonal treatment- estrogens or progestins.
4. Immunosuppressive/immunomodulating medication

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cell population | Through study completion, an average of 1 year
  The wash samples are processed, supernatant discarded and RBCs removed. Cells are then washed with FACS buffer ,subjected to antibody staining and examined by flow cytometry. Antibodies include: CD45,UV,CD3,CD19,CD66B,CD88, CD89, CD14,CD16,CD314,HLA-DR in order to identify monocytes, dendritic cells, T cells, B cells, NK and Neutrophil populations

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel